CLINICAL TRIAL: NCT03071289
Title: Observation Versus Radiation on Pelvic Lymphocysts After Radical Hysterectomy of Cervical Cancer: A Phase 3 Prospective Multi-institutional Randomised Controlled Trial
Brief Title: A Trial Comparing Observation With Radiation on Pelvic Lymphocysts After Radical Hysterectomy of Cervical Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei-jun Ye, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N2016203
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Cervical Cancer; Lymphocyst; Radiation Therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Lymphocele | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Group A) (Active Comparator): In Group A, adjuvant radio-chemotherapy is applied. The radiotherapy is performed according to Radiation Method A. The regimen of chemotherapy is cisplatin 30mg/m2 every week.
  Interventions: Drug: Cisplatin; Radiation: Radiation Method A
- The experiment group (Group B) (Experimental): In Group B, adjuvant radio-chemotherapy is applied. The radiotherapy is performed according to Radiation Method B. The regimen of chemotherapy is cisplatin 30mg/m2 every week.
  Interventions: Radiation: Radiation Method B; Drug: Cisplatin

INTERVENTIONS:
Radiation: Radiation Method B — The gross tumor volume (GTV) is the residual lesion after radical resection and given a dose of 60Gy. The clinical target volume (CTV) is delineated according to the lymph drainage pathway and included all the lymphocyst. The CTV is given a dose of 45Gy.
  Arms: The experiment group (Group B)
Drug: Cisplatin — The regimen of chemotherapy is cisplatin 30mg/m2 every week.
Radiation: Radiation Method A — The gross tumor volume (GTV) is the residual lesion after radical resection and given a dose of 60Gy. The clinical target volume (CTV) is delineated according to the lymph drainage pathway and given a dose of 45Gy.
  Arms: The control group (Group A)

SUMMARY:
Cervical cancer of early stage is treated mainly by radical resection and (or) radiotherapy. And pelvic lymphocyst is one of the most common adverse events of radical resection. The aim of this study is to compare observation with radiation on pelvic lymphocyst of cervical cancer patients after radical resection, for incidence of adverse events and local recurrence rate.

DETAILED DESCRIPTION:
1. Background

   Cervical Cancer is one of the most common malignant tumors of Chinese females. The early stage diseases (Stage Ia, Ib and IIa1) is treated mainly by radical resection and (or) radiotherapy. And pelvic lymphocyst is one of the most common adverse events (incidence 18-35%) of radical resection. When adjuvant radiotherapy (ART) is performed, lymphocyst is included in the clinical target volume (CTV) with a dose of 45-50Gy, in most hospitals of China. However, there is no pathologic and clinical evidence that lymphocyst is associated with local recurrence. However, inclusion of lymphocyst might enlarge CTV and increase irradiation dose of organs at risk (OARs) such as small intestine and kidneys.
2. Objective

   The aim of this study is to compare observation with radiation on pelvic lymphocyst of cervical cancer patients after radical resection, for incidence of adverse events and local recurrence rate.
3. Patients and methods

A patient will be enrolled when patient have:

1. pathologically diagnosed cervical cancer;
2. Stage I-II diseases (FIGO system ver. 2014);
3. treated with radical resection;
4. need of ART according to NCCN guidelines ver. 2016v2.

Randomization is performed to divide the patients into the control group (Group A) and the experimental group (Group B). In Group A, the CTV includes all the lymphocyst. But in Group B, the CTV is delineated according to the lymph drainage pathway (not all the lymphocyst included). ART is performed with a dose of 60Gy to the gross tumor volume, and 45Gy to the CTV. Chemotherapy is given concurrently with cisplatin 30mg/m2 every week regimen. The Grade 3/4 adverse events (CTCAE criteria ver. 4.03) and the 5-year local-recurrence-free survival of the 2 groups are compared after 5-year follow-up with an interval of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological diagnosed cervical cancer and treated with radical resection
* Stage I-II diseases (FIGO system ver. 2014)
* Karnofsky Performance Scores ≥ 80 and expected survival ≥ 3 months
* Pelvic MRI or CT indicate existence of lymphocyst
* Need of adjuvant radiotherapy according to NCCN guidelines ver. 2016v2 (SEDLIS criteria)

Exclusion Criteria:

* Patients with distant metastasis before or during radiotherapy
* Severe dysfunction of heart, lung, liver, kidney or hematopoietic system
* Severe neurological, mental or endocrine diseases
* History of other malignancies
* Prior chemotherapy, radiotherapy or application of monoclonal antibodies
* Patients participated in clinical trials of other drugs within last 3 months
* Pregnant or lactating women
* Those who are considered by the researchers unsuitable to participate

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
5-year local-recurrence-free survival (5y-LRFS) | 5 years after the date of radiotherapy completion
  Percentage of patients in a treatment group who are alive without local recurrence for a 5-year period of follow-up after the date of radiotherapy completion

SECONDARY OUTCOMES:
Incidence of grade 3/4 adverse event | Once a week during therapy, up to 5 years after the date of radiotherapy completion
  Incidence of patients in a treatment group who manifest a specific adverse event (such as myelosuppression) of grade 3/4. Incidence is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) criteria ver. 4.03.
5-year overall survival (5y-OS) | 5 years after the date of radiotherapy completion
  Percentage of patients in a treatment group who are alive for a 5-year period of follow-up after the date of radiotherapy completion

CONTACTS AND LOCATIONS:
Overall Officials: Wei-jun Ye, M.D, Principal Investigator — Sun Yat-sen University
Locations (8):
- China (8):
  - Sun Yat-sen University Affiliated Foshan Hospital, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Hospital of of Guangdong Armed Police Corps, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - Xinjiang Medical University Affiliated Tumor Hospital, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No